CLINICAL TRIAL: NCT05979077
Title: Improving Quality of Care in Diabetes Clinic Through Patient-Entered Electronic Health Data?
Brief Title: Children's Hospital Academic Medical Organization (CHAMO) MyChart Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Ellen Goldbloom, Pedatric Endocrinologist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22/99X
Record Dates: First submitted 2023-04-24; First posted 2023-08-07 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyChart Questionnaire (Intervention Group) (Experimental): Participants within the intervention group will complete the patient-facing EHR-enabled MyChart® questionnaire.
  Interventions: Other: MyChart Questionnaire
- Standard Clinical Care (Control Group) (No Intervention): Participants within the control group will undergo standard clinical care with no study intervention.

INTERVENTIONS:
Other: MyChart Questionnaire — Prior to clinic visits, families completing the MyChart Questionnaire will enter details about their current management and visit goals, automatically populating their electronic health record for subsequent review/revision by the health care team before and during the visit, reallocating clinic time previously used for data acquisition to individual patient priorities
  Arms: MyChart Questionnaire (Intervention Group)

SUMMARY:
Evolving technology and clinical innovation have led to dramatic changes in the management of type 1 diabetes (T1D). These changes have led to a need to collect a growing number of details from families during their visits. As a result, much of the physician-patient visit is spent transferring information instead of focusing on diabetes care, contributing to increased time pressures in clinic and unmet needs for patients.

In response to this reality, the investigators have developed a tool that allows families to input their diabetes-related information into their physicians' electronic health record (EHR) documentation tool before their clinic visit, using a questionnaire administered via CHEO's secure patient portal (MyChart®). The investigators will evaluate the impact of an integrated electronic patient questionnaire, on quality of care (patient-reported), diabetes control and clinic efficiency. The investigators hope that our study will determine whether having families input clinical data prior to a visit is an effective strategy to improve the quality of diabetes care. The investigators believe that the findings will be of interest to all those studying the value of incorporating patient-entered data both within diabetes care and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1D
* Age <11 years at enrollment

Exclusion Criteria:

* Patients ≥ 11 years of age at enrollment
* Patients who are not fluent enough in English to complete all study related procedures
* Patients unable or unwilling to provide consent and/or assent
* Patients followed in Eating Disorder Clinic or Child and Youth Protection Clinic (there are MyChart activation restrictions for individuals followed in these clinics)

Ages: 0 Years to 131 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of a patient-facing EHR-enabled questionnaire on patient-perceived quality of care. | 12 months
  The EHR-enabled questionnaire will be completed through the online MyChart portal. Patients' parents are required to complete diabetes-related questions across a total of 10 pages, including questions regarding the visit, insulin dosing, injection dose, insulin delivery, blood sugar monitoring, high blood glucose and ketones, hypoglycemia, nutrition, physical activity, and general health. These questions are typically addressed during routine clinic visits; however, they will be completed prior to the clinic visit and automatically entered into the patient's medical chart.
Patients' Evaluation of Quality of Diabetes Care (PEQD) | 12 months
  The PEQD is a brief and validated questionnaire designed to assess the participants' judgement about the quality of their diabetes care. It is scored on a scale of 0-100 with 100 representing the best possible quality of care.
Perceived Quality of Medical Care (PQMC) | 12 months
  The PQMC is a validated instrument designed to provide a simple, general measure of patients' overall quality of medical care they receive. Alpha reliability estimates should be expected to be above .90 for this instrument. It is scored on a scale from 6-42, with lower scores representing better perceived quality of medical care.
Participant Tool and Workflow Survey | 12 months
  This study-specific questionnaire was developed during pilot work for this study and was designed to specifically assess the myChart questionnaire being completed before each clinic visit. This questionnaire will only be given to those participants randomized to the intervention group. While this questionnaire has not been validated, it has been used in previously published research by our study team.

SECONDARY OUTCOMES:
To evaluate the impact of a patient-facing EHR-enabled questionnaire on glycemic control and visit efficiency. | 12 months
  Changes in glycemic control will be obtained from the patient's medical chart. Glycemic control will include: hemoglobin A1c (HbA1c, (%)), percent time in range (TIR - percentage of time in previous 14 days spent within target glucose range of 70-180 mg/dL or 3.9-10 mmol/L), and glucose management indicator (GMI, %).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Eastern Ontario - Research Institute, Ottawa, Ontario, Canada

DOCUMENTS (1):
  • Informed Consent Form (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT05979077/ICF_000.pdf